CLINICAL TRIAL: NCT05304481
Title: A Phase II Study to Evaluate the Efficacy and Safety of Activated T Lymphocytes (ATL) in Hepatocellular Carcinoma (HCC) Patients After Curative Treatment
Brief Title: Efficacy and Safety of Activated T Lymphocytes (ATL) in Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lukas Biomedical Inc. (Industry)
Collaborators: Virginia Contract Research Organization Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUKACTZ20171215
Record Dates: First submitted 2022-01-12; First posted 2022-03-31 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Oncology; Hepatocellular Carcinoma; Activated T lymphocytes
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): ATL administration
  Interventions: Biological: ATL administration

INTERVENTIONS:
Biological: ATL administration — Subjects have ATL administration using intravenous infusion

SUMMARY:
This is an open-label, single arm, multicenter, Phase II clinical study to investigate the efficacy and safety profiles of autologous ATL administration in HCC patients after curative treatment. Among all the eligible patients, ratio of 7:2:1 for Stage I:II:IIIa of the HCC will be the enrolled strategy of the study to reflect the results of the previous study (Lee, Lee et al. 2015).

DETAILED DESCRIPTION:
Eligible patients with HCC received curative treatment will be given ATL administration in this study. The investigational product ATL revealed great efficacy in previous clinical trials. This study aims to treat eligible patients, who had undergone curative treatment for HCC, with ATL as a preventive immunotherapy and to evaluate the effectiveness on the basis of patients' RFS rate in 12 months. The administration of the subject will be in a staggered manner for the first 3 patients. The 2nd and 3rd subject will not be dosed until the prior subject has taken the 4th dose of investigational products for at least 4 weeks. During the pretreatment period, peripheral blood for manufacturing the individualized ATL agent will be collected from patients at least 28 days before starting treatment. Patients will receive 200 mL of the ATL agent intravenously within 40 to 60 minutes without any premedication. They will be scheduled to receive the ATL 10 times at Weeks 1, 2, 3, 4, 6, 8, 10, 14, 18, and 22. A Data and Safety Monitoring Board (DSMB) will be appointed while 10% of schedule subjects were enrolled and complete 4 times of ATL infusions, the DSMB will convene a meeting to review safety data to date, including AEs and toxicities to indicate whether the study would advance unaltered, amend the protocol, or halt recruitment until a resolution of a specific issue.

ELIGIBILITY:
Inclusion Criteria for Donor

1. Patients must be able to understand and sign the informed consent documents and aware of the investigational nature of the study.
2. Patient is ≥ 20 years old.
3. Patient has been diagnosed as HCC by pathological data or radiological test in the stage of I, II or IIIa according to the American Joint Committee on Cancer staging system (8th Edition).
4. Patient is scheduled to or has received tumor removal by curative treatments (e.g., surgical operation, percutaneous ethanol injection [PEI], microwave ablation [MWA], or radiofrequency ablation [RFA]).
5. Patient meets below conditions by blood test, kidney and liver function test:

   White blood cell (WBC) count > 3,000/μL Absolute neutrophil count (ANC) ≥ 1,500/μL Hemoglobin (Hb) ≥ 9.0 g/dL Thrombocyte count > 50,000/μL Blood urea nitrogen (BUN) and serum Creatinine ≤ 1.5× Upper Limit of Normal (ULN) AST and ALT ≤ 5×ULN
6. Female patient with childbearing potential should be confirmed of not being pregnant at the screening and during the study.

Exclusion Criteria for Donor

1. Patient with syphilis, human immunodeficiency virus I/II (HIV-I/II), human T-lymphotropic virus I/II (HTLV-I/II), or an increased risk (or has been diagnosed) for human transmissible spongiform encephalopathy (TSE); including Creutzfeldt-Jakob disease (CJD)
2. Patient with ongoing active hepatitis including acute or active chronic HBV/HCV infection, alcohol-associated hepatitis, and autoimmune hepatitis, etc., according to site-specific diagnostic criteria and laboratory parameters at screening
3. Patient who has clinically significant and unstable gastrointestinal, renal, endocrine, pulmonary, or cardiovascular disease judged by the investigator
4. Patient who has disease history of malignancy other than HCC except for curatively treated non-melanoma skin cancer, cervical carcinoma in situ, or superficial bladder tumors within 5 years before participating in this clinical trial
5. Patient who has medical history of immune deficiency or auto-immune disease (including but not limited to: rheumatoid arthritis , Burger's disease, multiple sclerosis and Type I diabetes)
6. Patient with the following medication or treatment should be excluded as the donor:

   1. Systemic corticosteroids within 4 weeks prior to blood collection
   2. Immunosuppressive treatment within 4 weeks prior to blood collection
   3. Other anti-cancer treatments within 3 months prior to blood collection
   4. Attenuated vaccines within 4 weeks prior to blood collection
7. Patient who has participated in other investigational studies and received any investigational therapy within 4 weeks prior to blood collection
8. Patient who has known or suspected hypersensitivity to any ingredient in the product (e.g. kanamycin, streptomycin or albumin, etc.)

Inclusion Criteria for subject

1. Patient must be able to understand and has signed the informed consent documents and been aware of the investigational nature of the study.
2. Patient who has the histopathological or cytological proof (e.g. liver biopsy test) of HCC in the stage of I, II or IIIa. Patient's tumor has been totally removed by curative treatment (surgical operation, PEI, MWA or RFA) in 12 weeks based on the agreement date for written consent and the tumor's removal should be perfectly confirmed by medical imaging (Computed tomography (CT) scan or Magnetic resonance imaging (MRI)) within 4 weeks of first dosing.
3. Hepatic function of Child-Pugh class A
4. ECOG Performance status (ECOG-PS) score ≤ 1
5. Patient's remaining life-time is expected at least more than 3 months.
6. Patient meets below conditions by blood test, kidney and liver function test:

   WBC count > 3,000/μL ANC ≥ 1,500/μL Hb ≥ 9.0 g/dL Thrombocyte count > 50,000/μL BUN and serum Creatinine ≤ 1.5× ULN AST and ALT ≤ 5×ULN
7. Female patient with childbearing potential should be confirmed of not being pregnant or not lactating at the screening and during the study.
8. Patient is willing to comply with protocol-stated requirements, instructions and restrictions.
9. All male and female patients with child-bearing potential (between puberty and 2 years after menopause) are willing to use at least any one of the appropriate contraception methods shown below, for during and at least 24 weeks after ATL treatment.

   1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception).
   2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   3. Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
   4. Combination of any two of the following listed methods: (d.1+d.2 or d.1+d.3, or d.2+d.3):

   d.1Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

   d.2Placement of an intrauterine device (IUD) or intrauterine system (IUS). d.3Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps).

Exclusion Criteria for Subjects

1. Patient who has clinically significant and unstable gastrointestinal, renal, endocrine, pulmonary, or cardiovascular disease judged by the investigator
2. Patient with ongoing active hepatitis including acute or active chronic HBV/HCV infection, alcohol-associated hepatitis, and autoimmune hepatitis, etc., according to site-specific diagnostic criteria and laboratory parameters at screening.
3. Patient who has known or suspected hypersensitivity to any ingredient in the product (e.g. kanamycin, streptomycin or albumin, etc.)
4. Patient with the following medication or treatment should be excluded:

   1. Systemic corticosteroids within 4 weeks prior to receiving ATL or are scheduled to do so during the study.
   2. Immunosuppressive treatment within 4 weeks prior to receiving ATL or are scheduled to do so during the study.
   3. Other anti-cancer treatment within 4 weeks except for curative treatment prior to receiving ATL or are scheduled to do so during the study.
   4. Attenuated vaccines within 4 weeks prior to administration or is scheduled to do so during the study
5. Patient who fails to provide blood collection as a self-donor whose blood collection sample fails to generate adequate amount of ATL
6. Patient who is not able to take MRI or CT scan examination
7. Patient who has serious mental, social or psychological factors that may interfere with compliance and assessments of the study in the investigator's opinion
8. Patient who has participated in other investigational studies and received any investigational therapy within 4 weeks prior to the study dosing.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2022-05-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival rate | the baseline (the first dosing) to 12 months later from post-treatment
  the Relapse-free survival rate of ATL treated HCC patients

SECONDARY OUTCOMES:
Relapse-free survival | up to 76 weeks
  the time from baseline (the first dosing) to the first recurrence or death from any cause
Overall survival | up to 76 weeks
  the time from baseline (the first dosing) to death from any cause
Cancer-specific survival | Up to 24 months (estimated according to the average survival time)
  the time from baseline (the first dosing) to death resulting from HCC
Change of biomarkers | up to 76 weeks
  α-fetoprotein (AFP) and Protein Induced by Vitamin K Absence or Antagonist-II (PIVKA-II) level
Change in Eastern Cooperative Oncology Group (ECOG) performance status (for evaluation of change in the functional status) | up to 76 weeks
  Assessment with Eastern Cooperative Oncology Group (ECOG) score, in a range from 0 to 5 representing a status from better to worse.
Change in European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire score (for evaluation of quality of life) | up to 76 weeks
  Assessment with European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 version 3.0, while a higher score means a worse outcome.
Number of Participants With Abnormal Laboratory Values | up to 76 weeks
  Number of Participants who encounter abnormal lab test results which are clinically meaningful.
Change in body weight from baseline | up to 76 weeks
  body weight
AE incidences | up to 76 weeks
  Adverse event incidences
Number of Participants With Abnormal physical examination result | up to 76 weeks
  Number of Participants who encounter abnormal physical examination results which are clinically meaningful.
Change in ECG examination results | up to 76 weeks
  PR, QRS, QT, QTc, and RR intervals
Changes in body temperature | up to 76 weeks
  measurements of vital sign: body temperature
Changes in pulse rate | up to 76 weeks
  measurements of vital sign: pulse rate
Changes in blood pressures | up to 76 weeks
  measurements of vital sign: blood pressures including both systolic and diastolic pressure.
Changes in respiratory rate | up to 76 weeks
  measurements of vital sign: respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: Eric Tang, M.D., Study Director — Lukas Biomedical Inc.
Locations (13):
- Taiwan (13):
  - Hualien Tzu Chi Hospital, Hualien City, Taiwan
  - Cardinal Tien Hospital, New Taipei City, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan
  - Taipei City Hospital, RENAI Branch, Taipei, Taiwan
  - E-Da Cancer Treatment Hospital, Kaohsiung City
  - Far Estern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - Taipei Medical University Hospital, Taipei
  - Shin Kong Wu Ho Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No